CLINICAL TRIAL: NCT05770869
Title: mHealth ALIBIRD: A Digital Health Care Model (Analysis of the Applicability of an m-Health Platform and Its Impact on the Follow-up of Patients With Cancer: Pilot Study in a Sample of Patients With Advanced Non-small Cell Carcinoma)
Brief Title: mHealth ALIBIRD: A Digital Health Care Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Investigación E Innovación Biomédica Hospital Universitario Infanta Sofia-Henares (Other)
Collaborators: Hospital Infanta Sofia (Other); Universidad Politecnica de Madrid (Other); IMDEA Food (Other); Instituto de Investigación en Ciencias de la Alimentación (CIAL) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mHA
Record Dates: First submitted 2023-01-24; First posted 2023-03-16 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Thoracic Neoplasms
Keywords: Active Treatment
MeSH Terms: conditions — Thoracic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALIBIRD mHealth platform (Experimental): Participants are followed-up using the ALIBIRD mHealth platform. The ALIBIRD platform is made up of a mobile application for patients and a web application for the healthcare team. Through the ALIBIRD mobile application, patients regularly register Patients Reported Outcomes (PROs) and Patients Reported Outcome Measures (PROMs) regarding lifestyle (diet, physical activity, sleep, mood), and get access to individualized recommendations in order to assume more responsibility for achieving the best outcomes from their care. Moreover, the patient application includes features for tracking the appearance of symptoms, with alerts sent to the healthcare team in response to these parameters. In addition, the application contains articles and educational information.
  Interventions: Device: ALIBIRD mHealth platform

INTERVENTIONS:
Device: ALIBIRD mHealth platform — Use of a mHealth platform to follow-up and empower cancer patients in the self-management of their own health.

SUMMARY:
The aim of this pilot study was to evaluate the feasibility and acceptability of the ALIBIRD platform, a new mobile health (mHealth) application prototype design for personalized and remote support on the follow-up of cancer patients. The ALIBIRD platform is a mHealth intervention that tracks PROs, improving symptom control and allowing real-time feedback, and provides personalized recommendations and educational content, promoting empowerment and encourage healthy lifestyle behaviors in patients with thoracic neoplasms in active treatment.

DETAILED DESCRIPTION:
The investigators have developed an innovative mHealth platform that provides personalized recommendations based on Patient Reported Outcomes (PROs) records and the study of patient´s nutrigenomics and gut microbiome. The usability of the ALIBIRD mHealth platform prototype is being tested in a 28-week pilot study carried out at Infanta Sofía Hospital. A small group of stage IV thoracic neoplasms patients (n=20) were asked to participate. All the participants gave informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with thoracic neoplasms, histologically or cytologically confirmed.
* < 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patients receiving cancer treatment: chemotherapy, chemotherapy-immunotherapy, immunotherapy or biological therapy.
* Patients with internet access and intermediate level in the use of technology (Smartphone, mobile applications, wearable)
* Signed informed consent.

Exclusion Criteria:

* Patients with symptomatic brain metastases.
* Patients with neurological impairment, dementia or psychiatric disorders.
* Patients unable to follow the protocol due to psychological, social or geographic reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Usability and feasibility assesment | week 1 to 28
  Changes in Satisfaction System Usability Scale (SUS)

SECONDARY OUTCOMES:
Changes in Mediterranean Diet Serving Score (MDSS) | Week 1 to 28
  Mediterranean adherence assesment
Changes in Quality of life ( European Quality of Life-5 Dimensions 5 Levels questionnaire,EQ-5D-5L) from baseline | Week 1 to 28
  Quality of life assesment. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  In the VAS the individual scores his or her health between two extremes, 0 and 100, the worst and best state of health imaginable.
Changes in physical activity (International Physical Activity Questionnaire,PAQ) | Week 1 to 28
  Physical activity assesment
Changes in sleep (Pittsburg questionnaire) | Week 1 to 28
  Sleep assesment
Changes in Quality of life ( The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13, EORTC QLQ-LC-13) | Week 1 to 28
  Quality of life assesment. The LC13 covers 13 typical symptoms of lung cancer patients, such as coughing, pain, dyspnea, sore mouth, peripheral neuropathy, and hair loss. questions along 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning) and nine symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) All items are scored from 1 to 4 in relation to the presence of the symptom: not at all, a little, quite a bit, very much.
Changes in toxicity (Patient-Reported Outcome version of the Common Terminology Criteria for Adverse Events, PRO-CTAE questionnaire) | week 1 to 28
  Toxicity assesment
Changes is Hospital Anxiety and Depression Questionnaire (HADs) from baseline | Week 1 to 28
  Emotional status assesment. This is a scale containing two subscales with 7 anxiety symptoms (HADS-A) and 7 depression symptoms (HADS-D).
  The items are scored on a 4-point Likert frequency scale (0-3) with a total score ranging from 0 to 21 for each subscale, where a higher score is indicative of greater symptom severity.
Changes in Massachusetts General Hospital-Sexual Functioning Questionnaire (MGH-SFQ) from baseline | Week 1 to 28
  Sexuality assesment
Changes is medication adherence (MMAS-8 questionnaire) | Week 1 to 28
  Medication adherence assesment
Changes in belief in medication (Beliefs about Medicines Questionnaire,BMQ) | Week 1 to 28
  Belief in medication assesment

CONTACTS AND LOCATIONS:
Overall Officials: María Sereno Moyano, Medicine, Principal Investigator — Fundación Investigación E Innovación Biomédica Hospital Universitario Infanta Sofia-Henares
Locations (1):
- Servicio de Oncología. Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid, Spain